CLINICAL TRIAL: NCT00640913
Title: Early Reversal of Defunctioning Stoma Trial
Acronym: ELSOR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rectal Cancer Trial on Defunctioning Stoma Study Group (Other)
Responsible Party: Peter Matthiessen, MD, PhD, Department of Surgery, Örebro University Hospital, 701 85 Örebro
Other Study IDs: Ö 109-07
Record Dates: First submitted 2008-03-10; First posted 2008-03-21 (Estimated); Last update posted 2008-03-21 (Estimated); Status verified 2008-03

CONDITIONS: Rectal Cancer
Keywords: Defunctioning stoma; Low anterior resection; TME surgery; Early stoma reversal
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Analysis of serum C-Reactive Protein (CRP) and Procalcitonin (PCT).
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- I: Twenty consecutive patients operated on with low anterior resection of the rectum for cancer with a defunctioning stoma who accept participation.
  Interventions: Procedure: Reversal of defunctioning stoma

INTERVENTIONS:
Procedure: Reversal of defunctioning stoma — Reversal of defunctioning stoma

SUMMARY:
In this trial will be investigated if a defunctioning loop stoma used in low anterior resection of the rectum for cancer can be reversed after 14 days instead of 3-12 months which is present clinical practise.

DETAILED DESCRIPTION:
Patients undergoing low anterior resection of the the rectum for adenocarcinom (total mesorectal excision; TME) with a defunctioning loop stoma are assessed preoperatively and for 6 days postoperatively according to a trial protocol including daily clinical, physiological, and serological variables, and a rectal contrast study on day 6. If inclusion criteria are fulfilled, a decision is taken on day 7 to schedule reversal of the defunctioning loop stoma on postoperative day 14. This trial is considered a hypothesis generating pilot study of feasibility type and is no power calculation. The present trial will include 20 consecutive patients who accept participation.

ELIGIBILITY:
Inclusion Criteria:

* Written consent and fulfilled inclusion criteria preoperatively and during postoperative day 1-6.

Exclusion Criteria:

* Written consent and/or inclusion criteria not fulfilled preoperatively and during postoperative day 1-6.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty patients operated on with low anterior resection of the rectum for cancer and a defunctioning loop stoma.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-04 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Reversal of defunctioning loop stoma on postoperative day 14 following low anterior resection of the rectum for cancer with or without preoperative adjuvant treatment | Preoperatively, postoperative day 7, postoperative day 30 and at 6 months postoperatively

SECONDARY OUTCOMES:
Postoperative 30 day morbidity. Postoperative ano-rectal function at 1 and 6 months. | Postoperatively at 1 and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Matthiessen, MD, PhD, Principal Investigator — Department of Surgery, Örebro University Hospital
Locations (1):
- Department of Surgery, Örebro University Hospital, Örebro, Sweden